CLINICAL TRIAL: NCT01174160
Title: A Phase III, Prospective, Randomized, Double-Blind, Placebo-Controlled Multicenter Study to Evaluate the Efficacy and Safety of MK-6621 in Patients With Atrial Fibrillation
Brief Title: A Study of the Efficacy and Safety of Vernakalant Hydrochloride (MK-6621) in Patients With Atrial Fibrillation (MK-6621-010 AM4)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advanz Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6621-010
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vernakalant HCl (Experimental): vernakalant hydrochloride
  Interventions: Drug: vernakalant hydrochloride
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo to vernakalent hydrochloride

INTERVENTIONS:
Drug: vernakalant hydrochloride — Patients will receive a 3 mg/kg infusion of vernakalant hydrochloride. If the patient is in atrial fibrillation (AF) or atrial flutter (AFL) 25 minutes after the start of the infusion, then a second infusion of 2 mg/kg vernakalant hydrochloride will be administered.
  Other Names: MK-6621
  Arms: vernakalant HCl
Drug: Placebo to vernakalent hydrochloride — Patients will receive an infusion of placebo. If the patient is in atrial fibrillation (AF) or atrial flutter (AFL) 25 minutes after the start of the infusion, then a second infusion of placebo will be administered.
  Other Names: Saline
  Arms: placebo

SUMMARY:
This study will investigate if treatment with vernakalant hydrochloride (MK-6621) results in a greater proportion of patients with treatment-induced conversion of Atrial Fibrillation to sinus rhythm compared to placebo.

DETAILED DESCRIPTION:
Amendment 4 of the protocol revised the planned enrollment to 123 participants and removed China as one of the countries participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Abstinent or willing to use 2 acceptable methods of birth control
* Patient has an atrial arrhythmia with dysrhythmic symptoms
* Patient is receiving adequate anticoagulant therapy
* Patient has stable blood pressure
* Patient weighs between 45 and 136 kg (99 and 300 lbs)
* Patient is adequately hydrated

Exclusion Criteria:

* Patient is pregnant, breast-feeding, or expecting to become pregnant during the study
* Patient routinely consumes more than 2 alcoholic drinks per day
* Patient has known or suspected prolonged QT, familial long QT syndrome, previous Torsades de Pointes, Brugada syndrome
* Patient has known bradycardia, advanced AV block, or sick-sinus syndrome, unless controlled by a pacemaker
* Patient has severe aortic stenosis
* Patient has atrial flutter
* Patient has Class IV congestive heart failure (CHF)
* Patient has had a myocardial infarction (MI) or acute coronary syndrome (ACS)
* Patient has had cardiac surgery within 30 days
* Patient has known atrial thrombus
* Patient has reversible causes of Atrial Fibrillation
* Patient has failed electrical cardioversion during current episode of Atrial Fibrillation
* Patient has uncorrected electrolyte imbalance
* Patient has clinical evidence of digoxin toxicity
* Patient has received certain antiarrhythmic drugs or intravenous amiodarone within 7 days
* Patient is known to be HIV positive
* Patient has a history of cancer within the past 5 years, except for certain skin or cervical cancers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Vernakalant IV: vernakalant hydrochloride
  Up to two 10-min infusions of 3mg/kg +/- 2mg/kg vernakalant IV
- Placebo: placebo
  Up to two 10-min infusions of normal saline
Period: Overall Study
Arm/Group | Vernakalant IV | Placebo
Started | 61 | 62
Discontinued Pre Dose | 6 | 6
Dosed | 55 | 56
Discontinued Post Dose | 2 | 0
Completed | 53 | 56
Not Completed | 8 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 4 | 6
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vernakalant IV | Placebo | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (13.7) | 59.2 (12.0) | 59.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 26 | 44
  Male | 37 | 30 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 54 | 56 | 110
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 55 | 55 | 110
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 42 | 48 | 90
  India | 0 | 1 | 1
  Taiwan | 13 | 7 | 20
New York Heart Association (NYHA) Classification [Number; unit: participants] — NHYA classifies the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina pain.
  participants
    None (no heart failure) | 50 | 53 | 103
    Class I (cardiac disease but no symptoms) | 1 | 1 | 2
    Class II (mild symptoms during normal activity) | 2 | 2 | 4
    Class III (Marked limitation in activity) | 2 | 0 | 2
Structural Heart Disease [Number; unit: participants] — Participants could have been classified in more than one category
  participants
    None | 44 | 43 | 87
    Congestive Heart Failure | 5 | 3 | 8
    Ischemic Heart Disease | 4 | 7 | 11
    Myocardial Infarction | 1 | 0 | 1
    Valvular Heart Disease | 2 | 3 | 5
Atrial fibrillation (AF) duration [Number; unit: participants]
  Less than or equal to 48 hours | 33 | 31 | 64
  More than 48 hours | 22 | 25 | 47

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Treatment-induced Conversion of Atrial Fibrillation to Sinus Rhythm
Description: The proportion of patients with treatment-induced conversion of atrial fibrillation to sinus rhythm for a minimum duration of 1 minute
Time Frame: Within 90 minutes after first exposure
Measure: Number; unit: participants
Arm/Group | Vernakalant IV | Placebo
Number analyzed (Participants) | 55 | 56
participants | 29 | 7

ADVERSE EVENTS:
Arm/Group | Vernakalant IV | Placebo
Serious Adverse Events (participants affected / at risk) | 6/55 | 6/56
Other Adverse Events (participants affected / at risk) | 23/55 | 23/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vernakalant IV (N=55) | Placebo (N=56)
Arrhythmia (Cardiac disorders) | 1 | 0
Congestive Heart Failure (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 0 | 2 — General disorders and administration site conditions
Cerebral infarction (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1
Acute renal failure (Renal and urinary disorders) | 1 | 0
Neurogenic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vernakalant IV (N=55) | Placebo (N=56)
Bradycardia (Cardiac disorders) | 4 | 2
Ventricular tachycardia (Cardiac disorders) | 1 | 4
Sick sinus syndrom (Cardiac disorders) | 2 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Wound complications (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Acute renal failure (Renal and urinary disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to submit a copy of a 'Publication' to CRO/Sponsor for review and comment 60 days prior to submission for publication and / or disclosure. Sponsor has the applicable 60 day period to respond to PI with any requested revisions. PI agrees to delete any confidential information (excluding results) identified by Sponsor as confidential prior to submitting/presenting the publication.